CLINICAL TRIAL: NCT06700720
Title: A Phase Ⅱa Clinical Study to Evaluate the Efficacy and Safety of YN001 in Patients With Coronary Atherosclerosis in Australia
Brief Title: YN001-004 in Patients With Coronary Atherosclerosis in Australia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Beijing Inno Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YN001-004
Record Dates: First submitted 2024-11-14; First posted 2024-11-22 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-04

CONDITIONS: Coronary Artery Disease; Coronary Atherosclerotic Disease
Keywords: Coronary Atherosclerosis; Plaque regression
MeSH Terms: conditions — Coronary Artery Disease | interventions — evolocumab

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dose 1 treatment arm (Experimental): Dose 1 YN001 will be administrated intravenously weekly.
  Interventions: Drug: Dose 1 YN001; Drug: Evolocumab
- Dose 2 treatment arm (Experimental): Dose 2 YN001 will be administrated intravenously weekly.
  Interventions: Drug: Dose 2 YN001; Drug: Evolocumab

INTERVENTIONS:
Drug: Dose 1 YN001 — Dose 1 YN001 will be administered on Day 1 of each week from Week 1 to Week 13, 13 times in total.
  Arms: Dose 1 treatment arm
Drug: Dose 2 YN001 — Dose 2 YN001 will be administered on Day 1 of each week from Week 1 to Week 13, 13 times in total.
  Arms: Dose 2 treatment arm
Drug: Evolocumab — Evolocumab 140 mg will be administered subcutaneously every 2 weeks.
  Other Names: Repatha®

SUMMARY:
This study is to evaluate the efficacy and safety of intravenously administered YN001 in patients with coronary atherosclerosis in Australia. This study will be conducted in eligible participants with a diagnosis of coronary atherosclerosis, and at least 1 coronary artery is blocked determined by coronary computed tomography angiography (CCTA)

DETAILED DESCRIPTION:
This is a multicenter, randomized, open label, parallel-group, proof of concept study. It is designed to determine if the study drug, called YN001, administered in addition to evolocumab can effectively reduce the total amount of plaque formed in the coronary artery as measured by CCTA from baseline to week 13.

A total of 24 patients with coronary atherosclerosis are expected to be enrolled and will be randomly assigned in a 1:1 ratio to 1 of 2 YN001 treatment arms (12 patients per arm) with 2 different dose levels for 12 weeks.

The study will be comprised of a maximum 41-day screening period (Day -42-Day -2), a baseline period (Day-1), a treatment and observation period (W1D1- W13D7), and a safety follow-up period (14 days post last dose).

ELIGIBILITY:
Inclusion Criteria:

1. Fully understand the purposes, features, and methods of the study, and sign the ICF before performing any assessment.
2. Male or female Australia patients between 18 and 75 years.
3. Patients diagnosed with coronary atherosclerosis, and at least 1 vessel with diameter stenosis determined by coronary computed tomography angiography (CTA).
4. Female patients must be non-pregnant and non-lactating, and females of childbearing potential (including a female partner of a male patient) must agree to use 1 effective contraception method from the screening period to 3 months after receiving their last dose of the study drug. In addition, male patients must be willing to refrain from sperm donation during this time.
5. Willing and able to comply with the requirements of protocol to the best of the patient's and investigator's knowledge.

Exclusion Criteria:

1. Prior treatment with other investigational drug(s) within 30 days or 5 half-lives, whichever is longer, prior to randomization.
2. Previously received YN001.
3. Any type of vaccination within 4 weeks prior to randomization.
4. Contraindication for coronary CTA (e.g., known history of anaphylactic contrast reactions).
5. Multi-vessel severe disease.
6. Recent acute ST-segment elevation myocardial infarction (STEMI) occurred within 2 weeks prior to randomization.
7. Relapse and highly symptomatic arrhythmia uncontrolled by drugs within the past 3 months, such as ventricular tachycardia, atrial fibrillation with rapid ventricular rate and paroxysmal supraventricular tachycardia.
8. Prior treatment with CABG, heart transplantation, SAVR/TAVR, etc., or CABG, heart transplantation, SAVR/TAVR, etc., is required or planned during the study.
9. PCI performed within 4 weeks prior to randomization or PCI is required or planned during study treatment.
10. New York Heart Association (NYHA) class III or IV, or last known left ventricular ejection fraction (LVEF) <40%.
11. Recent clinically evident stroke occurred within 6 months prior to randomization (except for TIA).
12. Presenting with history of myopathy/myalgia, or susceptible to myopathy/rhabdomyolysis.
13. Known inflammatory bowel disease, ulcers, gastrointestinal or rectal bleeding within 6 months prior to randomization.
14. Evidence of major diseases that not recovered within 2 weeks prior to randomization, or major surgery is expected during the study.
15. Presenting with history of malignancy (except in patients who have been disease-free >5 years; or whose only malignancy has been basal or squamous cell skin carcinoma).
16. Presence of any type of autoimmune disease.
17. Allergy to multiple food or drugs or known sensitivity to any components to be administered during dosing
18. Life expectancy is less than 1 year.
19. Systolic blood pressure of ≥150 mmHg at final screening despite antihypertensive therapy.
20. Known familial hypercholesterolemia
21. Triglycerides≥400 mg/dl (4.5 mmol/l) at final screening.
22. Active liver disease or hepatic dysfunction defined by any of ALT, AST, or total bilirubin > 2 times upper limit of normal (ULN) at final screening.
23. Presence of renal insufficiency.
24. Untreated or inadequately treated hypothyroidism defined by thyroid stimulating hormone (TSH) > 1.5 times ULN at final screening.
25. Poorly controlled (defined by HbA1c > 9%) type 2 diabetes mellitus.
26. A positive hepatitis B surface antigen (HBsAg), or positive antibody against hepatitis C virus (anti-HCV) or human immunodeficiency virus (anti-HIV), or positive treponema pallidum antibody (TP-Ab).
27. Current smoker who has smoked an average of≥5 cigarettes (or equivalent) per day over the preceding year.
28. Presence of any other diseases or conditions (apart from those outlined above) that, in the opinion of the investigator, would make it unsuitable for the patient to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Changes in coronary plaque characteristics (volume and composition) | From baseline to Week 13
  Evaluating YN001 on top of evolocumab therapy in changing coronary plaque volume assessed by coronary computed tomography angiography (CCTA).

SECONDARY OUTCOMES:
Change in mean of mean carotid IMT | From baseline to Week 13
  Evaluating YN001 on top of evolocumab therapy in changing carotid intima-media thickness (IMT) assessed by carotid ultrasound.
Change in mean of mean carotid IMT | From baseline to Week 5
  Evaluating YN001 on top of evolocumab therapy in changing carotid intima-media thickness (IMT) assessed by carotid ultrasound.
Change in mean of mean carotid IMT | From baseline to Week 9
  Evaluating YN001 on top of evolocumab therapy in changing carotid intima-media thickness (IMT) assessed by carotid ultrasound.
Change in mean peri-coronary Fat attenuation index (FAI) | From baseline to Week 13
  Evaluating YN001 on top of evolocumab therapy in changing inflammation using the peri-coronary FAI value measured by quantitative CTA analysis.
The safety profile of YN001 | From baseline to Week 15
  Incidence of Adverse events (AEs)/Serious adverse events (SAEs)
Plasma concentration of total and free drug | From Week 1 to Week 13
  Plasma concentration of total and free drug at pre-dose (0 h) and at the end of infusion
Population pharmacokinetics (PK) | From Week 1 to Week 13
  Plasma PK parameter (AUC) and patient covariates of interest will be evaluated graphically and in the population PK model.

OTHER OUTCOMES:
Immunogenicity（ADA） analysis | From Week 1 to Week 13
  The proportion of patients who develop anti-drug antibodies (ADA) following drug administration.
Immunogenicity （APA）analysis | From screening to Week 13
  The proportion of patients with pre-exsiting anti-PEG antibodies (APA), treatment emergent APA or treatment boosted APA following drug administration.
Exploratory dose-response analysis of plaque volume | From Week 1 to Week 13
  Exploratory dose-response analysis will be performed by comparing the difference of coronary plaque volume changing between 2 different dose levels
Exploratory dose-response analysis of AEs | From Week 1 to Week 13
  Exploratory dose-response analysis will be performed by comparing the difference of incidence of AEs between 2 different dose levels

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Chen, PhD, Study Director — Beijing Inno Medicine Co., Ltd.
Locations (6):
- Australia (6):
  - Canberra Hospital, Canberra, Australian Capital Territory
  - Albury Wodonga Private Hospital, Albury, New South Wales
  - Sunshine Coast University Private Hospital, Birtinya, Queensland
  - Core Research Group Pty Ltd, Milton, Queesland
  - Altona Clinical Research, Melbourne, Victoria
  - Peninsula Heart Centre, Melbourne, Victoria